

## STATISTICAL ANALYSIS PLAN

Study Title: A Phase 2 Randomized, Open Label, Active Controlled Study

Evaluating the Safety and Efficacy of Long-acting Capsid Inhibitor GS-6207 in Combination with Other Antiretroviral

Agents in People Living with HIV

Name of Test Drug: Lenacapavir (LEN; GS-6207)

Study Number: GS-US-200-4334

Protocol Version (Date): Amendment 4 (04 February 2022)

Analysis Type: Final Analysis

Analysis Plan Version: Version 1.0

Analysis Plan Date: 17 January 2024

Analysis Plan Author(s): PPD

CONFIDENTIAL AND PROPRIETARY INFORMATION

## TABLE OF CONTENTS

| TΑ | BLE O | F CONTE | NTS | 2 |
|---|---|---|---|---|
| LIS | T OF I | N-TEXT T | 'ABLES | 4 |
| | | | ATIONS | |
| PH | ARMA | RMACOKINETIC ABBREVIATIONS | | |
| 1. | INTR | ODUCTIO | ON | 8 |
| | 1.1. | Study O | Objectives | 9 |
| | 1.2. | | esign | |
| | 1.3. | | Size and Power | |
| 2. | TVP | - | NNED ANALYSIS | |
| 2. | | | | |
| | 2.1. | | Analyses | |
| | | 2.1.1. | DMC Analysis | |
| | | 2.1.2.<br>2.1.3. | Week 28 Interim Analysis | |
| | 2.2 | | Week 80 Interim Analysis | |
| | 2.2.<br>2.3. | | Analysis | |
| 3. | GEN | ERAL CO | NSIDERATIONS FOR DATA ANALYSES | 13 |
| | 3.1. | Analysis | s Sets | 13 |
| | | 3.1.1. | | |
| | | 3.1.2. | | |
| | | 3.1.3. | Safety Analysis Set | 13 |
| | | 3.1.4. | Pharmacokinetic Analysis Set | 14 |
| | 3.2. | | ant Grouping | |
| | 3.3. | | nd Covariates | |
| | 3.4. | Examin | ation of Participant Subgroups | |
| | | 3.4.1. | | |
| | 3.5. | | e Comparisons | |
| | 3.6. | | Data and Outliers | |
| | | 3.6.1. | 0 | |
| | | 3.6.2. | | |
| | 3.7. | | andling Conventions and Transformations | |
| | 3.8. | | s Visit Windows | |
| | | 3.8.1. | | |
| | | 3.8.2. | Analysis Visit Windows | 18 |
| | | 3.8.3. | Selection of Data in the Event of Multiple Records in an Analysis Visit Window | 10 |
| , | DAD | TICIDANIT | DISPOSITION | |
| 4. | | | | |
| | 4.1. | | ant Enrollment and Disposition | |
| | 4.2. | | rug Administration and Adherence | |
| | | 4.2.1. | Study Drug Administration | |
| | | 4.2.2. | Study Drug Adherence | |
| | | | 4.2.2.1. Adherence to SC LEN | |
| | 4.2 | Ch. 4. D | 4.2.2.2. Adherence to Once Daily Study Drug(s) | |
| | 4.3.<br>4.4. | | Puration | |
| | 4.4. | FIGUCO | I Deviations | 23 |
| 5 | BASI | FLINE CH | ARACTERISTICS | 26 |

| | 5.1.<br>5.2. | | aphics and Baseline Characteristics aseline Characteristics | |
|---|---|---|---|---|
| | 5.3. | | History | |
| 6. | EFFICACY ANALYSES | | | |
| | 6.1. | 6.1. Primary Efficacy Endpoint | | |
| | 6.2. | Secondary Efficacy Endpoints | | |
| | | 6.2.1. | Definition of the Secondary Efficacy Endpoints | |
| | | 6.2.2. | Primary Analysis for the Secondary Endpoints | |
| | | 6.2.3. | Secondary Analysis for the Secondary Endpoints | |
| | CCI | | | |
| | 6.4. | Changes | s from Protocol-Specified Efficacy Analysis | 29 |
| 7. | SAFE | SAFETY ANALYSES | | |
| | 7.1. | Adverse | Events and Deaths | 30 |
| | | 7.1.1. | Adverse Event Dictionary | |
| | | 7.1.2. | Adverse Event Severity | |
| | | 7.1.3. | Relationship of Adverse Events to Study Drug | |
| | | 7.1.4. | Serious Adverse Events | |
| | | 7.1.5. | Treatment-Emergent Adverse Events. | |
| | | 6.5 (C) (C) (C) | 7.1.5.1. Definition of Treatment-Emergent Adverse Events | |
| | | | 7.1.5.2. Incomplete Dates | |
| | | 7.1.6. | Summaries of Adverse Events and Deaths. | |
| | | /.1.0. | 7.1.6.1. Summaries of AE incidence in Combined Severity Grade | |
| | | | Subsets | 31 |
| | | 7.1.7. | Additional Analysis of Adverse Events | |
| | | 7.1.7. | 7.1.7.1. Study Drug Related Injection Site Reactions | |
| | | | 7.1.7.2. Study Drug Related Injection Site Reactions 7.1.7.2. Study Drug Related Injection Site Induration and Nodules | |
| | 7.2. | Laborate | ory Evaluations | |
| | 1.4. | 7.2.1. | Summaries of Numeric Laboratory Results | |
| | | 7.2.2. | Graded Laboratory Values | |
| | | 1.4.4. | 7.2.2.1. Treatment-Emergent Laboratory Abnormalities | |
| | | | 7.2.2.1. Summaries of Laboratory Abnormalities | |
| | 7.3. | D. J. W | /eight and Vital Signs | |
| | 7.4. Prior and Concomitant Medications | | | |
| | | 7.4.1. | Nonstudy Drug Antiretroviral Medications | |
| | | 7.4.2. | Concomitant Non-ARV Medications | |
| | 7.5. | 7.5.1 | ardiogram Results | |
| | 20 | | Investigator Electrocardiogram Assessment | |
| | 7.6. | Other Safety Measures Participant Subgroup for Safety Endpoints | | |
| | 7.7. | Changes From Protocol-Specified Safety Analysis | | |
| 0 | 7.8. | | | |
| 8. | PHARMACOKINETIC (PK) ANALYSES | | | |
| | 8.1. | 1 1 つきままします。 これは 1 つきまました 1 つきまま 1 つきまま 1 つきまま 2 つきま 2 つき 2 つき | | |
| | 8.2. | | lyses Related to PK Sampling. | |
| | | 8.2.1. | Statistical Analysis Methods | |
| | | 8.2.2. | Sensative Analysis | |
| | 8.3. | | | |
| 9. | | EFERENCES | | |
| 10. | SOFT | SOFTWARE | | |

| 11. | SAP REVISION | | 44 |
|---|---|---|---|
| 12. | APPENDICES | | 45 |
| | | LIST OF IN-TEXT TABLES | |
| | Table 3-1. | Analysis Visit Windows for HIV-1 RNA, CD4+ cell count, CD4 %, Hematology, Chemistry, Lipid Panel, Urinalysis, Urine Chemistry, Urine Pregnancy Laboratory Tests, Vital Signs, and Weight for the LEN-containing Regimen Groups (Treatment Groups 1-3) | 18 |
| | Table 3-2. | Analysis Visit Windows for HIV-1 RNA, CD4+ cell count, CD4 %, Hematology, Chemistry, Lipid Panel, Urinalysis, Urine Chemistry, Urine Pregnancy Laboratory Tests, Vital Signs, and Weight for the B/F/TAF Group (Treatment Group 4) | |

#### LIST OF ABBREVIATIONS

AE adverse event

ALT alanine aminotransferase
AST aspartate aminotransferase
BLQ below the limit of quantitation

BMI body mass index

CFR Code of Federal Regulations

CI confidence interval
CK creatine kinase
CRF case report form
CSR clinical study report

CTCAE Common Terminology Criteria for Adverse Events

DILI drug-induced liver injury
DMC data monitoring committee

ECG electrocardiogram
ET early termination
FAS Full Analysis Set
Hb hemoglobin
HLT high-level term

ICH International Conference on Harmonization (of Technical Requirements for Registration of

Pharmaceuticals for Human Use)

ITT intent to treat
LTT lower-level term
LOQ limit of quantitation

MedDRA Medical Dictionary for Regulatory Activities

PP per protocol PT preferred term

Q1, Q3 first quartile, third quartile

QRS electrocardiographic deflection between the beginning of the Q wave and termination of the

S wave representing time for ventricular depolarization

QT electrocardiographic interval between the beginning of the Q wave and termination of the

T wave representing the time for both ventricular depolarization and repolarization to occur

QTc QT interval corrected for heart rate

QTcF QT interval corrected for heart rate using Fridericia's formula

RR electrocardiographic interval representing the time measurement between the R wave of one

heartbeat and the R wave of the preceding heartbeat

SAP statistical analysis plan SD standard deviation

SI (units) international system of units

SOC system organ class

| TEAE | treatment-emergent adverse event |
|------|----------------------------------|
| TFLs | tables, figures, and listings |
| ULN | upper limit of normal |
| VR | ventricular rate |
| WHO | World Health Organization |

#### PHARMACOKINETIC ABBREVIATIONS

AUC<sub>last</sub> area under the concentration versus time curve from time zero to the last quantifiable

concentration

AUCtau area under the concentration versus time curve over the dosing interval

Clast last observed quantifiable concentration of the drug

C<sub>max</sub> maximum observed concentration of drug

C<sub>tau</sub> observed drug concentration at the end of the dosing interval CLss/F apparent oral clearance after administration of the drug:

at steady state: CLss/F = Dose/AUCtau, where "Dose" is the dose of the drug

t<sub>1/2</sub> estimate of the terminal elimination half-life of the drug, calculated by dividing the natural log of

2 by the terminal elimination rate constant ( $\lambda_z$ )

 $T_{last}$  time (observed time point) of  $C_{last}$   $T_{max}$  time (observed time point) of  $C_{max}$ 

λz terminal elimination rate constant, estimated by linear regression of the terminal elimination

phase of the concentration of drug versus time curve

#### 1. INTRODUCTION

This statistical analysis plan (SAP) describes the statistical analysis methods and data presentations to be used in tables, figures, and listings (TFLs) in the clinical study report (CSR) for Study GS-US-200-4334. This SAP is based on the study protocol amendment 4 dated 04 February 2022 and the electronic case report form (eCRF). The SAP will be finalized before database finalization. Any changes made after the finalization of the SAP will be documented in the CSR.

## 1.1. Study Objectives

The primary objective of this study is as follows:

 To evaluate the efficacy of LEN containing regimens in people living with HIV (PLWH) as determined by the proportion of participants with HIV-1 RNA < 50 copies/mL at Week 54</li>

The secondary objectives of this study are as follows:

- To evaluate the efficacy of LEN containing regimens in PLWH as determined by the proportion of participants with HIV-1 RNA < 50 copies/mL at Weeks 28, 38, and 80</li>
- To evaluate the change from baseline in log<sub>10</sub> HIV-1 RNA and in CD4+ cell count at Weeks 28, 38, 54, and 80
- To evaluate the safety and tolerability of the LEN containing regimens through 28, 38, 54, and 80 weeks of treatment
- To evaluate the pharmacokinetics (PK) of LEN, bictegravir (BIC), and tenofovir alafenamide (TAF)

## 1.2. Study Design

## **Design Configuration and Participant Population**

This is a Phase 2, randomized, open label, active controlled, multicenter study.

Approximately 175 treatment-naive PWH who meet all eligibility criteria will be randomized in a 2:2:2:1 ratio to 1 of the following 4 treatment groups. Randomization will be stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening.

## Treatment Groups

## Treatment Group 1 (n = 50)

Induction: Participants will receive oral LEN 600 mg, 600 mg, and 300 mg, without regard to food, at Days 1, 2, and 8 respectively. Participants will also begin oral daily emtricitabine (F)/TAF (200/25 mg), without regard to food from Day 1 onwards for a total of 28 weeks. On Day 15 participants will receive subcutaneous (SC) LEN 927 mg, without regard to food.

Maintenance: Participants will receive SC LEN 927 mg at Week 28 and every 26 weeks thereafter. Participants will discontinue oral daily F/TAF (200/25 mg) at Week 28 and begin taking oral daily TAF (25 mg), without regard to food.

### Treatment Group 2 (n = 50)

Induction: Participants will receive oral LEN 600 mg, 600 mg, and 300 mg, without regard to food at Days 1, 2, and 8 respectively. Participants will also begin oral daily F/TAF (200/25 mg), without regard to food from Day 1 onward for a total of 28 weeks. On Day 15 participants will receive SC LEN 927 mg, without regard to food.

Maintenance: Participants will receive SC LEN 927 mg at Week 28 and every 26 weeks thereafter. Participants will discontinue oral daily F/TAF (200/25 mg) at Week 28 and begin oral daily BIC (75 mg) without regard to food.

## Treatment Group 3 (n = 50)

Participants will receive oral LEN 600 mg and 600 mg without regard to food at Days 1 and 2, respectively. On Day 3, participants will begin oral daily LEN 50 mg, without regards to food. Participants will begin oral daily F/TAF (200/25 mg), without regard to food from Day 1 onwards.

#### Treatment Group 4 (n = 25)

Participants will receive oral daily bictegravir/emtricitabine/TAF (B/F/TAF, 50/200/25 mg), without regard to food at Day 1 and throughout their participation in the study.

#### Key Eligibility Criteria

Treatment naive PWH who meet the following criteria:

- Age ≥ 18 years of age at Screening
- Plasma HIV-1 RNA ≥ 200 copies/mL at Screening
- CD4+ cell count ≥ 200 cells/µL at Screening
- Antiretroviral (ARV) naive with no use of any ARV medications within one month of Screening. Use of pre-exposure prophylaxis (PrEP) (any duration), post-exposure prophylaxis (PEP) (any duration), or HIV-1 treatment (< 10 days therapy total) > 1 month prior to Screening is permitted.

#### Schedule of Assessments

At screening, laboratory analyses (hematology, chemistry, and urinalysis, and serum pregnancy test [for women]), HIV-1 RNA, CD4+ cell count, vital signs, electrocardiogram (ECG), complete physical examination and estimated glomerular filtration rate (eGFR) will be performed, and hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies will be analyzed. Analysis of the participant's HIV-1 resistance to support eligibility will be completed.

After screening procedures, eligible participants will be randomized into 1 of the 4 treatment groups in a 2:2:2:1 ratio.

Participants in Treatment Groups 1, 2, and 3 only, will have visits on Day 1, Day 2, CCI, Day 8, and Day 15. All participants will have a Week 4 visit and will continue to attend study visits every 6 weeks until Week 28.

Participants in Treatment Groups 1 and 2 will need to have HIV-1 RNA results < 50 copies/mL at Weeks 16 and 22 to initiate treatment with a two agent regimen at Week 28; those with values > 50 copies/mL will discontinue the study drug at or prior to Week 28.

After Week 28, participants will attend study visits on Week 38, Week 54, Week 64, and Week 80. After Week 80, participants in Treatment Group 4 will complete the study and participants in Treatment Groups 1, 2, and 3 will be given the option to receive further treatment and continue to attend visits alternating between every 10 weeks and every 16 weeks visits.

At each visit, adverse events (AEs), concomitant medications, laboratory tests, physical examinations, PK, and patient reported outcomes (PROs) will be performed in accordance with the Study Procedures Table.

More details for study procedures could be found in Section 12 (Appendix 1).

#### Study Duration

Duration of treatment is at least 80 weeks. Participants in Treatment Group 4 will complete the study at Week 80.

Following successful completion of Week 80 visit, participants receiving LEN will be given the option to receive further treatment and continue to attend visits on Week 90, Week 106, Week 116, Week 132, Week 142, and will continue to alternate between every 10 weeks and every 16 weeks visits. Participants willing to continue the study beyond Week 80 in Treatment Groups 1 and 2 will continue to receive SC LEN 927 mg every 6 months (26 weeks) from Week 80 onwards and participants in Treatment Group 3 will receive oral LEN 50 mg daily from Week 80 until the product becomes accessible to participants through an access program, or until Gilead elects to discontinue the study in the country. Participants in Treatment Groups 1, 2, and 3 will also receive TAF, F/TAF, or BIC as applicable.

Participants who discontinue study drugs prior to Week 80 visit or prior to study completion may be required to complete 30-Day, 90-Day and/or 180-Day Follow Up visits after Early Termination Visit.

## Oral Weekly Bridging of LEN for Missed SC Injection

Participants receiving SC LEN may miss their SC injection window (within 26 to 28 weeks of the previous SC LEN dose). If a missed dose is anticipated, participants may receive oral bridging until they can receive their next SC injection.

## 1.3. Sample Size and Power

A sample size of 50 participants in Treatment Groups 1 to 3, respectively, was chosen to estimate the response rate of HIV-1 RNA < 50 copies/mL at Week 54. A total sample size of 75 participants for each pair of comparisons (ie, between each of the LEN-containing regimen groups [Treatment Groups 1 to 3, n = 50] and the B/F/TAF [Treatment group 4, n = 25]) will provide 39% power to evaluate non-inferiority with respect to the response rate of HIV-1 RNA < 50 copies/mL at Week 54. In this sample size and power calculation, it is assumed a response rate is 90.9% (based on pooled data from Studies GS-US-380-1489 and GS-US-380-1490) for each treatment group and a non-inferiority margin is 0.12.

#### 2. TYPE OF PLANNED ANALYSIS

## 2.1. Interim Analyses

#### 2.1.1. DMC Analysis

One external multidisciplinary Data Monitoring Committee (DMC) analysis was conducted after all participants have completed their Week 16 visit or prematurely discontinued from study drug, all outstanding data queries had been resolved or adjudicated as unresolvable, and the data had been cleaned and finalized for the analysis. No formal stopping rules was used by the DMC for safety outcomes. Rather, a clinical assessment was made to determine if the nature, frequency, and severity of AEs associated with a study treatment warrant the early termination of the study in the best interest of the participants. No alpha penalty will be applied for the primary analysis of the primary efficacy endpoint given that the study is not adequately powered for a formal efficacy evaluation. The purpose of the interim analysis was to provide the DMC with a statistical report for review. More details are documented in the DMC charter.

#### 2.1.2. Week 28 Interim Analysis

The Week 28 interim analysis was conducted after all participants have completed the Week 28 visit or have prematurely discontinued the study drug, outstanding data queries had been resolved or adjudicated as unresolvable, and the data had been cleaned and finalized for the analysis. The analysis was used to support the LEN regulatory filing for the indication in the heavily treatment experienced PWH.

### 2.1.3. Week 80 Interim Analysis

The Week 80 interim analysis was conducted after all participants have completed the Week 80 visit or have prematurely discontinued the study drug, outstanding data queries had been resolved or adjudicated as unresolvable, and the data had been cleaned and finalized for the analysis.

## 2.2. Primary Analysis

The Week 54 interim analysis was conducted after all participants have completed Week 54 visit or have prematurely discontinued the study drug, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized for the analysis. This is the primary analysis of this study.

## 2.3. Final Analysis

The final analysis will be performed after all participants have completed the study, outstanding data queries have been resolved or adjudicated as unresolvable, and the data have been cleaned and finalized.

This SAP describes the analysis plan for the Final Analysis.

#### 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

Analysis results will be presented using descriptive statistics. For categorical variables, the number and percentage of participants in each category will be presented; for continuous variables, the number of participants (n), mean, standard deviation (SD) or standard error (SE), median, first quartile (Q1), third quartile (Q3), minimum, and maximum will be presented.

All statistical tests will be 2-sided and performed at the 5% significance level unless otherwise specified.

By-participant listings will be presented for all participants in the All Randomized Analysis Set and sorted by participant ID number, visit date, and time (if applicable). Data collected on log forms, such as AEs, will be presented in chronological order within the participant. The treatment group to which participants were randomized will be used in the listings. Age, sex at birth, race, and ethnicity will be included in the listings, as space permits.

#### 3.1. Analysis Sets

Analysis sets define the participants to be included in an analysis. Analysis sets and their definitions are provided in this section. The analysis set will be identified and included as a subtitle of each table, figure, and listing.

For each analysis set, the number and percentage of participants eligible for inclusion will be summarized by treatment group.

A listing of reasons for exclusion from analysis sets will be provided by participant.

## 3.1.1. All Randomized Analysis Set

All Randomized Analysis Set includes all participants who were randomized in the study.

This is the primary analysis set for by-participant listings.

#### 3.1.2. Full Analysis Set

The Full Analysis Set (FAS) includes all randomized participants who took at least 1 dose of study drug. This is the primary analysis set for efficacy analyses.

## 3.1.3. Safety Analysis Set

The Safety Analysis Set includes all participants who took at least 1 dose of study drug. This is the primary analysis set for safety analyses.

#### 3.1.4. Pharmacokinetic Analysis Set

The Pharmacokinetic (PK) Analysis Set will include all randomized participants who took at least 1 dose of study drug and have at least 1 nonmissing concentration value reported by the PK laboratory. This is the primary analysis set for all PK analyses.

## 3.2. Participant Grouping

For analyses based on the All Randomized Analysis Set or the FAS, participants will be grouped according to the treatment group to which they were randomized. For all other analyses, participants will be grouped according to the actual treatment received. The actual treatment received will differ from the randomized treatment only when their actual treatment differs from randomized treatment for the entire treatment duration.

Participants will be grouped as follows for table summary:

- Treatment Group 1: SC LEN + (F/TAF → TAF)
- Treatment Group 2: SC LEN + (F/TAF → BIC)
- Treatment Group 3: Oral LEN + F/TAF
- Treatment Group 4: B/F/TAF
- Treatment Groups 1 and 2: SC LEN (for all tables unless specified otherwise)
- Treatment Groups 1, 2, and 3: LEN (for all tables unless specified)

#### 3.3. Strata and Covariates

Randomization was stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening.

Efficacy analyses will include HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) at baseline as a stratification factor. The HIV-1 RNA stratum will be reclassified using baseline HIV-1 RNA level for analysis purposes.

#### 3.4. Examination of Participant Subgroups

#### 3.4.1. Participant Subgroups for Safety Analyses

Incidence of all treatment-emergent AEs (TEAEs) will be analyzed for the following participant subgroups:

- Age (years): (a) < 50 and (b) ≥ 50</li>
- Sex: (a) male and (b) female
- Race: (a) black and (b) nonblack

## 3.5. Multiple Comparisons

Adjustments for multiplicity will not be made in this Phase 2, non-confirmatory trial.

## 3.6. Missing Data and Outliers

## 3.6.1. Missing Data

In general, missing data will not be imputed unless methods for handling missing data are specified. Exceptions are presented in this document.

For missing last dosing date of study drug, imputation rules are described in Section 3.8.1. The handling of missing or incomplete dates for AE onset is described in Section 7.1.5.2, and for prior and concomitant medications in Section 7.4.

#### 3.6.2. Outliers

Outliers will be identified during the data management and data analysis process, but no sensitivity analyses will be conducted. All data will be included in the data analysis.

## 3.7. Data Handling Conventions and Transformations

Only year of birth is collected in this study. The following conventions will be used for the imputation of date of birth when it is partially missing or not collected:

- If only month and year of birth is collected, then "15" will be imputed as the day of birth
- If only year of birth is collected, then "01 July" will be imputed as the day and month of birth
- If year of birth is missing, then date of birth will not be imputed.

In general, age collected at Day 1 (in years) will be used for analyses and presented in listings. If age at Day 1 is not available for a participant, then age derived based on date of birth and the Day 1 visit date will be used instead. If an enrolled participant was not dosed with any study drug, the randomization date will be used instead of the Day 1 visit date. For screen failures, the date the first informed consent was signed will be used for the age derivation. Age required for longitudinal and temporal calculations and analyses (eg, estimates of creatinine clearance, age at date of AE) will be based on age derived from date of birth and the date of the measurement or event, unless otherwise specified.

Non-PK data that are continuous in nature but are less than the lower limit of quantitation (LOQ) or above the upper LOQ will be imputed as follows:

- A value that is 1 unit less than the lower LOQ at the same precision level of the originally reported value will be used to calculate descriptive statistics if the datum is reported in the form of "< x" (where x is considered the lower LOQ). For example, if the values are reported as < 50 and < 5.0, values of 49 and 4.9, respectively, will be used to calculate summary statistics. An exception to this rule is any value reported as < 1 or < 0.1, etc. For values reported as < 1 or < 0.1, a value of 0.9 or 0.09, respectively, will be used to calculate summary statistics.</p>
- A value that is 1 unit above the upper LOQ will be used to calculate descriptive statistics if
  the datum is reported in the form of "> x" (where x is considered the upper LOQ). Values
  with decimal points will follow the same logic as above.
- The lower or upper LOQ will be used to calculate descriptive statistics if the datum is reported in the form of "≤x" or "≥x" (where x is considered the lower or upper LOQ, respectively).

Sparse PK concentration values that are below the limit of quantitation (BLQ) will be presented as "BLQ" in the data listing.

Logarithmic (base 10) transformations will be applied to HIV-1 RNA data for efficacy analysis. HIV-1 RNA results of "No HIV-1 RNA detected" and "<20 cp/mL HIV-1 RNA Detected" will be imputed as 19 copies/mL for analysis purposes.

Natural logarithm transformation will be used for analyzing concentrations and PK parameters in intensive PK samples. Concentration values that are BLQ will be presented as "BLQ" in the concentration data listing. Values that are BLQ will be treated as 0 at predose time points, and one-half the value of the LOQ at postdose time points for summary purposes.

The following conventions will be used for the presentation of summary and order statistics for intensive PK concentrations:

- If at least 1 participant has a concentration value of BLQ for the time point, the minimum value will be displayed as "BLQ."
- If more than 25% of the participants have a concentration data value of BLQ for a given time point, the minimum and Q1 values will be displayed as "BLQ."
- If more than 50% of the participants have a concentration data value of BLQ for a given time point, the minimum, Q1, and median values will be displayed as "BLQ."
- If more than 75% of the participants have a concentration data value of BLQ for a given time point, the minimum, Q1, median, and Q3 values will be displayed as "BLQ."
- If all participants have concentration data values of BLQ for a given time point, all order statistics (minimum, Q1, median, Q3, and maximum) will be displayed as "BLQ."

PK parameters that are BLQ will be imputed as one-half LOQ before log transformation or statistical model fitting.

#### 3.8. Analysis Visit Windows

## 3.8.1. Definition of Study Day

Study Day 1 is defined as the day when the first dose of study drug was taken, as recorded on the Study Drug Administration eCRF. For participants in Treatment Groups 1-3, the earliest of the first dose dates of any component (ie, LEN or F/TAF) is considered as the first dose date of the study drug.

Last Dose Date is defined as follows for participants who prematurely discontinued study drug in Treatment Groups 1 to 3, or completed study drug at main phase in Treatment Group 4 according to Study Drug Completion eCRF (ie, "study drug completion" box checked "No" for participants who prematurely discontinued, or "study drug completion" box checked "Yes" for participants who completed study drug in Treatment Group 4).

- For participants who receive SC injection, the last dose date is defined as the latest nonmissing end date of the study drug used with LEN.
- For participants who do not receive SC injection, the last dose date is defined as the earliest
  of the last dose date of any study drug.
- If the date of last dose is incomplete or missing (eg, due to lost to follow-up), the latest
  nonmissing study drug start dates and end dates, the clinic visit dates, and the laboratory visit
  dates excluding the dates of any follow-up visits will be used to impute the last dose date.

Study Days are calculated relative to Study Day 1 of study drug and derived as follows:

- For postdose study days: Assessment Date First Dose Date + 1
- For days prior to the first dose: Assessment Date First Dose Date

Baseline Value is defined as the last value obtained on or prior to the first dose of study drug.

Last Study Date is the latest nonmissing clinic visit dates, and/or the laboratory visit dates, and/or latest AE onset date and end date, whichever is latest, including the any follow-up visit dates, for participants who prematurely discontinued study according to the Study Completion eCRF.

Last Exposure Date is defined as follows for participants who prematurely discontinued study drug according to Study Drug Completion eCRF. This date is defined considering the prolonged exposure of LEN after the last dose date of LEN.

- Treatment Groups 1 and 2:
  - For participants who receive SC injection, last exposure date is defined as last study date.
  - For participants who do not receive SC injection, last exposure date is defined as the minimum of the last dose date plus 60 days and the last study date.

- Treatment Group 3: last exposure date is defined as the minimum of the last dose date plus 60 days and the last study date.
- Treatment Group 4: last exposure date is defined as the minimum of the last dose date plus 30 days and the last study date.

## 3.8.2. Analysis Visit Windows

Participant visits might not occur on protocol-specified days. Therefore, for the purpose of analysis, observations will be assigned to analysis windows.

The analysis windows for HIV-1 RNA, CD4+ cell count, CD4 %, hematology, chemistry, lipid panel, urinalysis, urine chemistry, urine pregnancy laboratory tests, vital signs, and weight are provided in Table 3-1 and Table 3-2 for the LEN-containing regimen groups (Treatment Groups 1-3) and the B/F/TAF group (Treatment Group 4), respectively.

Table 3-1. Analysis Visit Windows for HIV-1 RNA, CD4+ cell count, CD4 %, Hematology, Chemistry, Lipid Panel, Urinalysis, Urine Chemistry, Urine Pregnancy Laboratory Tests, Vital Signs, and Weight for the LEN-containing Regimen Groups (Treatment Groups 1-3)

| | | Visit Window Study Day | |
|----------|-----------|------------------------|-------------|
| Visit | Study Day | Lower Limit | Upper Limit |
| Day 1 | 1 | ≤1 | 1 |
| Day 2 | 2 | 2 | 5 |
| Day 8 | 8 | 6 | 11 |
| Day 15 | 15 | 12 | 21 |
| Week 4 | 28 | 22 | 49 |
| Week 10 | 70 | 50 | 91 |
| Week 16 | 112 | 92 | 133 |
| Week 22 | 154 | 134 | 175 |
| Week 28 | 196 | 176 | 231 |
| Week 38 | 266 | 232 | 322 |
| Week 54 | 378 | 323 | 413 |
| Week 64 | 448 | 414 | 504 |
| Week 80 | 560 | 505 | 595 |
| Week 90 | 630 | 596 | 686 |
| Week 106 | 742 | 687 | 777 |
| Week 116 | 812 | 778 | 868 |
| Week 132 | 924 | 869 | 959 |
| Week 142 | 994 | 960 | 1050 |
| Week 158 | 1106 | 1051 | 1141 |
| Week 168 | 1176 | 1142 | 1232 |
| Week 184 | 1288 | 1233 | ≥ 1288 |

Table 3-2. Analysis Visit Windows for HIV-1 RNA, CD4+ cell count, CD4 %, Hematology, Chemistry, Lipid Panel, Urinalysis, Urine Chemistry, Urine Pregnancy Laboratory Tests, Vital Signs, and Weight for the B/F/TAF Group (Treatment Group 4)

| | | Visit Window Study Day | |
|---------|-----------|------------------------|-------------|
| Visit | Study Day | Lower Limit | Upper Limit |
| Day 1 | 1 | ≤1 | 1 |
| Week 4 | 28 | 2 | 49 |
| Week 10 | 70 | 50 | 91 |
| Week 16 | 112 | 92 | 133 |
| Week 22 | 154 | 134 | 175 |
| Week 28 | 196 | 176 | 231 |
| Week 38 | 266 | 232 | 322 |
| Week 54 | 378 | 323 | 413 |
| Week 64 | 448 | 414 | 504 |
| Week 80 | 560 | 505 | ≥ 560 |

# 3.8.3. Selection of Data in the Event of Multiple Records in an Analysis Visit Window

Depending on the statistical analysis method, single values may be required for each analysis window. For example, change from baseline by visit usually requires a single value, whereas a time-to-event analysis would not require 1 value per analysis window.

If multiple valid, nonmissing measurements exist in an analysis window, records will be chosen based on the following rules if a single value is needed:

- For baseline, the last nonmissing value on or prior to the first dose date of study drug will be
  selected, unless specified differently. If there are multiple records with the same time or no
  time recorded on the same day, the baseline value will be the average of the measurements
  for continuous data (except for HIV-1 RNA, see below), or the measurement with the lowest
  severity (eg, normal will be selected over abnormal for safety ECG findings) for categorical
  data.
- For postbaseline values:
  - The record closest to the nominal day for that visit will be selected with the exception of CD4 cell counts and CD4% in which the latest record will be selected and HIV-1 RNA level (see below)
  - If there are 2 records that are equidistant from the nominal day, the later record will be selected.

- If there is more than 1 record on the selected day, the average will be taken for continuous data (except for HIV-1 RNA, see below) and the worse severity will be taken for categorical data, unless otherwise specified.
- For baseline and postbaseline HIV-1 RNA, the latest (considering both date and time) record(s) in the window will be selected. If both HIV test results ("HIV RNA Cobas 6800" or "HIV RNA Taqman 2.0") and repeated HIV test results ("HIV RNA Cobas6800RPT" or "HIV RNA Repeat", ie, the HIV-1 RNA result obtained from an additional aliquot of the original sample) are available with the same collection time, the results from the "HIV RNA Repeat" will be selected for analysis purposes; otherwise, if there are multiple "HIV RNA Cobas 6800" records with the same collection time, the geometric mean will be taken for analysis purposes.

#### 4. PARTICIPANT DISPOSITION

#### 4.1. Participant Enrollment and Disposition

Key study dates (ie, first participant screened, first participant randomized, last participant last visit for the primary endpoint, and last participant last visit for the clinical study report) will be provided.

A summary of participant enrollment will be provided by treatment group for each country, investigator within a country, and overall. The summary will present the number and percentage of participants randomized. For each column, the denominator for the percentage calculation will be the total number of participants analyzed for that column.

A similar enrollment table will be provided by randomization stratum. The denominator for the percentage of participants in the stratum will be the total number of randomized participants. If there are discrepancies in the value used for stratification assignment between the interactive web response system (IXRS) and the clinical database, the value collected in the clinical database will be used for the summary. A listing of participants with discrepancies in the value used for stratification assignment between the IXRS and the clinical database at the time of data finalization will be provided. If there are differences between randomization stratum using screening HIV-1 RNA value and baseline HIV-1 RNA value, a listing of the differences will also be provided.

The randomization schedule used for the study was provided as an appendix to the Week 28 CSR.

A summary of participant disposition will be provided by treatment group and total based on all screened participants. This summary will present the number of participants screened, the number of participants who met all eligibility criteria but were not randomized with reasons participants not randomized, the number of participants randomized but never dosed (if applicable), the number of participants randomized, and the number of participants in each of the categories listed below:

- Safety Analysis Set
- Continuing study drug in the main phase
- Completed study drug in the main phase
- Did not complete study drug with reasons for premature discontinuation of study drug in the main phase (if applicable)
- Completed study drug in the main phase and not entering the extension phase
- Completed study drug in the main phase and entering in the extension phase

- Entering and treated in the extension phase
- Continuing study drug in the extension phase
- Completed study drug in the extension phase
- Did not complete study drug with reasons for premature discontinuation of study drug in the extension phase (if applicable)
- Continuing study
- Completed study
- Did not complete the study with reasons for premature discontinuation of study (if applicable)

Duration of treatment is at least 80 weeks. At Week 80, participants in Treatment Group 4 will complete the study. Participants in Treatment Groups 1, 2, and 3 will be given the option to receive further treatment and continue to attend visits beyond Week 80. Main phase data is defined as the data collected on/before Week 80 visit. Extension phase data is defined as the data collected after Week 80 visit.

For the status of study drug and study completion and reasons for premature discontinuation, the number and percentage of participants in each category will be provided. The denominator for the percentage calculation will be the total number of participants in the Safety Analysis Set corresponding to that column in that study phase (if applicable). In addition, a flowchart will be provided to depict the disposition.

The following by-participant listings will be provided by participant ID number in ascending order to support the above summary tables:

- Reasons for premature study drug or study discontinuation
- Reasons for screen failure (will be provided by screening ID number in ascending order)

## 4.2. Study Drug Administration and Adherence

Study drug administration and study drug dispensing information will be collected in the Study Drug Administration and Study Drug Accountability eCRFs. All data including lot number and kit ID (if applicable) will be listed.

## 4.2.1. Study Drug Administration

Study drug administration and study drug dispensing information will be collected in the Study Drug Administration and Study Drug Accountability eCRFs. Number of participants receiving oral lead-in LEN and SC LEN at each protocol specified visit (Day 1, Day 2, for oral LEN and Day 15, Week 28, Week 54, Week 80, Week 106, and etc. for SC LEN) will be summarized.

Number of participants receiving oral reload before the first SC injection due to missed scheduled oral dosing, and number of participants receiving oral bridging after the first SC injection will also be provided.

## 4.2.2. Study Drug Adherence

Adherence to SC LEN and Once Daily Study Drug(s) will be derived except for oral lead-in LEN and oral bridging LEN in Treatment Groups 1 and 2.

#### 4.2.2.1. Adherence to SC LEN

The adherence to SC LEN will be assessed by adherence to the projected injection interval, which is 26 weeks (182 days) between 2 adjacent injection visits. The number of days from the projected injection visit date will be calculated for each injection visit (excluding the 1<sup>st</sup> injection visit) as the injection visit date minus the previous injection visit date minus 182 days minus oral bridging period (ie, First Dose Date of Resumed SC Injection - First Dose Date of Oral Bridging) if any occurred between these 2 adjacent injection visits. The number of days from the projected injection visit date will be classified into the following categories

- < -14 days</li>
- -14 to -8 days
- -7 to -3 days
- ± 2 days
- 3 to 7 days
- 8 to 14 days
- > 14 days

The number and percentage of participants in each category will be summarized for participants in Treatment Groups 1 and 2 who receive SC injections for the injection visit of interest.

## 4.2.2.2. Adherence to Once Daily Study Drug(s)

The adherence to once daily (QD) study drug(s) will be calculated based on 1 study drug for Treatment Groups 1, 2, and 4 (ie, F/TAF up to Week 28 and TAF or BIC from Week 28 onwards for Treatment Groups 1 and 2, and B/F/TAF for Treatment Group 4), and 2 study drugs for Treatment Group 3 (ie, oral QD LEN and F/TAF), excluding long acting LEN used for oral lead-in and oral bridging.

Adherence (%) of QD study drug(s) will be calculated as follows:

Adherence (%) = 
$$100 \times \frac{Total \text{ No. of pills taken}}{Total \text{ No. of pills prescribed}}$$

$$= 100 \times \frac{\sum \sum \text{No. of pills taken at each dispensing period for each study drug}^{[1]}}{\sum \sum \text{No. of pills prescribed at each dispensing period for each study drug}^{[2]}}$$

- [1] Number of pills taken at a distinct dispensing period for QD study drug(s) will be calculated as the minimum of (a) the daily number of pills prescribed multiplied by the duration of treatment of QD study drug(s) at the dispensing period of the same dispensing date, and (b) the number of pills taken (number of pills dispensed minus the number of pills returned). Total number of pills taken is determined by summing the number of pills taken from all evaluable dispensing periods for all QD study drug(s).
- [2] Number of pills prescribed at a distinct dispensing period for QD study drug(s) will be calculated as the daily number of pills prescribed multiplied by the duration of treatment of QD study drug(s) at the dispensing period of the same dispensing date. Total number of pills prescribed is determined by summing the number of pills prescribed from all evaluable dispensing periods for all QD study drug(s).

The duration of treatment of QD study drug(s) at a dispensing period for the study drug is calculated as the minimum of (a) the last returned date of the study drug at a dispensing period, (b) date of premature discontinuation of the study drug, and (c) next pill dispensing date of the study drug, minus dispensing date of the study drug.

The next pill dispensing date is the following dispensing date of the study drug regardless of the bottle return date.

For a record where the number of pills returned was missing (with "Yes" answered for "Was Bottle returned?" question), it is assumed the number of pills returned was zero. If the number of pills dispensed was missing or any study drug bottle was not returned or the bottle return status was unknown, all records in that dispensing period for that study drug will be excluded from both denominator and numerator calculation.

Adherence will be calculated for each participant for the entire dosing period up to the date of permanent discontinuation of the study drug for participants who prematurely discontinued study drug or using all available data for participants ongoing on study drug by the data cut date.

Descriptive statistics for adherence (n, mean, SD, median, Q1, Q3, minimum, and maximum) along with the number and percentage of participants belonging to adherence categories (eg,  $< 80\%, \ge 80\%$  to  $< 90\%, \ge 90\%$  to  $< 95\%, \ge 95\%$ ) will be provided for participants who return at least 1 bottle of randomized QD study drug, and who have calculable adherence in the Safety Analysis Set. No inferential statistics will be provided.

A by-participant listing of study drug administration and drug accountability will be provided separately by participant ID number (in ascending order) and visit (in chronological order).

## 4.3. Study Duration

Due to long acting feature of LEN, duration of follow-up to study drug will consider the prolonged exposure of LEN after the last dose date of LEN. Duration of exposure to study drug will be defined as (the last exposure date – the first dose date + 1), and will be expressed in weeks using up to 1 decimal place (eg, 4.5 weeks). Last exposure date is defined in Section 3.8.1 for participants who prematurely discontinued study drug.

Duration of exposure will be summarized using descriptive statistics (n, mean, SD, median, Q1, Q3, minimum, and maximum) and as the number and percentage of participants exposed and remained through the following time periods: 1 day, 2 days, 8 days, 15 days, 4 weeks (28 days), 10 weeks (70 days), 16 weeks (112 days), 22 weeks (154 days), 28 weeks (196 days), etc. Summaries will be provided based on the Safety Analysis Set. No inferential statistics will be provided.

#### 4.4. Protocol Deviations

Participants who did not meet the eligibility criteria for study entry but enrolled in the study, will be summarized regardless of whether they were exempted by the sponsor or not. The summary will present the number and percentage of participants who did not meet at least 1 eligibility criterion and the number of participants who did not meet specific criteria by treatment group based on the All Safety Analysis Set. A by-participant listing will be provided for those participants who did not meet at least 1 eligibility (inclusion or exclusion) criterion. The listing will present the eligibility criterion (or criteria if more than 1 deviation) that participants did not meet and related comments, if collected.

Protocol deviations occurring after participants entered the study are documented during routine monitoring. The number and percentage of participants with important protocol deviations (eg, at least 1, with 1, 2, 3 or more important protocol deviations), and the total number of important protocol deviations by deviation category (eg, eligibility criteria, informed consent) will be summarized by treatment group for the Safety Analysis Set. A by-participant listing will be provided for those participants with important protocol deviation.

#### 5. BASELINE CHARACTERISTICS

## 5.1. Demographics and Baseline Characteristics

Participant demographic variables (ie, age, sex at birth, gender identity, sexual orientation, race, and ethnicity) and baseline characteristics (body weight [in kg], height [in cm], body mass index [BMI; in kg/m²]) will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of participants for categorical variables. The summary of demographic data will be provided for the Safety Analysis Set.

Statistical comparison across treatment groups will be performed. For categorical data, the Cochran-Mantel-Haenszel (CMH) test will be used to compare across treatment groups except for gender identity and sexual orientation. For continuous data, the 2-sided Kruskal-Wallis test will be used to compare across treatment groups.

A by-participant demographic listing, including the informed consent date, will be provided by participant ID number in ascending order.

#### 5.2. Other Baseline Characteristics

The following baseline disease characteristics will be summarized by treatment group and overall using descriptive statistics for continuous variables and using number and percentage of participants for categorical variables:

- HIV-1 RNA (log<sub>10</sub> copies/mL)
- HIV-1 RNA categories (copies/mL): (a) ≤ 100,000, (b) > 100,000
- CD4 cell counts (/uL)
- CD4 cell counts categories (/uL): (a) < 50, (b) ≥ 50 to < 200, (c) ≥ 200 to < 350,</li>
   (d) ≥ 350 to < 500, and (e) ≥ 500</li>
- CD4 percentage (%)

The summary of these baseline disease characteristics will be provided for the Safety Analysis Set. Statistical comparison across treatment groups will be conducted similarly as described for the demographic and baseline characteristics.

A by-participant listing of other baseline characteristics will be provided by participant ID number in ascending order.

#### 5.3. Medical History

General medical history data will be collected at screening including HIV-1 disease-related events. General medical history data will be coded and listed.

#### 6. EFFICACY ANALYSES

## 6.1. Primary Efficacy Endpoint

The primary efficacy endpoint is the proportion of participants with HIV-1 RNA < 50 copies/mL at Week 54 as determined by the United States (US) Food and Drug Administration (FDA)-defined snapshot algorithm {U. S. Department of Health and Human Services 2015}. The proportions are expressed as percentages for presentation purposes.

The statistical analysis methods for the primary efficacy endpoint were described in the Week 54 SAP and the analysis was performed in the Week 54 analyses.

## 6.2. Secondary Efficacy Endpoints

## 6.2.1. Definition of the Secondary Efficacy Endpoints

The secondary efficacy endpoints of this study are:

- The proportion of participants with HIV-1 RNA < 50 copies/mL at Weeks 28, 38, and 80 as
  determined by the US FDA-defined snapshot algorithm</li>
- The change from baseline in log<sub>10</sub> HIV-1 RNA and in CD4+ cell count at Weeks 28, 38, 54, and 80

## 6.2.2. Primary Analysis for the Secondary Endpoints

The proportion of participants with HIV-1 RNA < 50 copies/mL at Weeks 28, 38, and 80 as determined by the US FDA-defined snapshot algorithm has been performed in the Weeks 28, 54, and Week 80 analyses and will not be repeated here.

## 6.2.3. Secondary Analysis for the Secondary Endpoints

The change from baseline in log<sub>10</sub> HIV-1 RNA and in CD4+ cell counts will be based on the FAS and summarized up to the visits with available data using descriptive statistics. The differences in changes from baseline in log<sub>10</sub> HIV-1 RNA and CD4+ cell count between each of the LEN-containing treatment groups (Treatment Groups 1-3) and the B/F/TAF group (Treatment Group 4) and the associated p-values and 95% CIs will be constructed using analysis of variance (ANOVA) models adjusting for the baseline HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL).

Mean  $\pm$  95% CI and median (Q1, Q3) of the change from baseline in  $log_{10}$  HIV-1 RNA and CD4+ cell counts will be plotted by visit

## 6.3. Other Efficacy Endpoints

# 6.3.1. Proportion of Participants with HIV-1 RNA < 50 copies/mL by Missing = Failure and Missing = Excluded Analyses

Number and percentage of participants with HIV-1 RNA < 50 copies/mL by visit will be analyzed using the following 2 analyses:

Missing = Failure (M = F):

In this approach, missing data will be treated as virologic failure and summarized into the "missing" category (see list of HIV-RNA categories below).

Missing = Excluded (M = E):

In this approach, missing data will be excluded in the computation of the percentages (ie, missing data points will be excluded from both the numerator and denominator in the computation). The denominator for percentages at a visit is the number of participants in the FAS with nonmissing HIV-1 RNA value at that visit.

For both M = F and M = E analyses, the number and percentage of participants with HIV-1 RNA in the following categories will be summarized based on the FAS:

- < 50 copies/mL</p>
  - < 20 copies/mL</p>
    - < 20 copies/mL Not Detectable</p>
    - < 20 copies/mL Detectable</p>
  - 20 to < 50 copies/mL</p>
- 50 to < 200 copies/mL</li>
- 200 to < 400 copies/mL</li>
- 400 to < 1000 copies/mL</li>
- ≥ 1000 copies/mL
- Missing (only applicable to M = F analysis)

Statistical comparison between each of the LEN-containing treatment groups (Treatment Groups 1-3) and the B/F/TAF group (Treatment Group 4) will be performed. Point estimates and its 95% CIs will be estimated using stratum-adjusted MH proportion as described in Section 6.2.3. The associated p-values will be estimated based on the CMH test stratified by baseline HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL).

## 6.4. Changes from Protocol-Specified Efficacy Analysis

No change from protocol-specified efficacy analysis is planned.

#### 7. SAFETY ANALYSES

Safety data will be summarized for participants in the Safety Analysis Set. All safety data collected up to the last exposure date for participants who prematurely discontinued study drug. All collected data will be included in data listings.

#### 7.1. Adverse Events and Deaths

## 7.1.1. Adverse Event Dictionary

Clinical and laboratory AEs will be coded using the current version of Medical Dictionary for Regulatory Activities (MedDRA). System organ class (SOC), high-level group term (HLGT), high-level term (HLT), preferred term (PT), and lower-level term (LLT) will be provided in the AE dataset.

## 7.1.2. Adverse Event Severity

Adverse events are graded by the investigator as Grade 1, 2, 3, 4, or 5 according to toxicity criteria specified in the protocol. The severity grade of events for which the investigator did not record severity will be categorized as "missing" for tabular summaries and data listings. The missing category will be listed last in summary presentation.

#### 7.1.3. Relationship of Adverse Events to Study Drug

Related AEs are those for which the investigator selected "Related" on the AE CRF to the question of "Related to Study Treatment." Relatedness will always default to the investigator's choice, not that of the medical monitor. Events for which the investigator did not record relationship to study drug will be considered related to study drug for summary purposes. However, by-participant data listings will show the relationship as missing.

## 7.1.4. Serious Adverse Events

Serious adverse events (SAEs) will be identified and captured as SAEs if the AEs met the definitions of SAEs that were specified in the study protocol. SAEs captured and stored in the clinical database will be reconciled with the SAE database from the Gilead Global Patient Safety (GLPS) Department before data finalization.

## 7.1.5. Treatment-Emergent Adverse Events

#### 7.1.5.1. Definition of Treatment-Emergent Adverse Events

Treatment-emergent adverse events (TEAEs) are defined as 1 or both of the following:

Any AEs leading to premature discontinuation of study drug, or

 Any AEs with an onset date on or after the study drug start date and no later than the last exposure date after permanent discontinuation of the study drug.

#### 7.1.5.2. Incomplete Dates

If the onset date of the AE is incomplete and the AE stop date is not prior to the first dose date of study drug, then the month and year (or year alone if month is not recorded) of onset determine whether an AE is treatment emergent. The event is considered treatment emergent as follows:

- Participants who receive SC injection: the AE onset date is the same as or after the month and year (or year) of the first dose date of study drug
- Participants who do not receive SC injection:
  - The AE onset is the same as or after the month and year (or year) of the first dose date of study drug, and
  - The AE onset date is the same as or before the month and year (or year) of the last exposure date

An AE with completely missing onset and stop dates, or with the onset date missing and a stop date later than the first dose date of study drug, will be considered to be treatment emergent. In addition, an AE with the onset date missing and incomplete stop date with the same or later month and year (or year alone if month is not recorded) as the first dose date of study drug will be considered treatment emergent.

When calculating the duration of event or time to onset, the following imputation rule will be used:

Missing start month/day: Jan 1/first day of the month will be used unless this is before the start date of study drug; in this case the study drug start date will be used;

Missing stop month/day: Dec 31/last day of the month will be used, unless this is after the last study date; in this case the last study date will be used.

Completely missing start or end dates will remain missing, with no imputation applied.

#### 7.1.6. Summaries of Adverse Events and Deaths

Treatment-emergent AEs will be summarized based on the Safety Analysis Set.

#### 7.1.6.1. Summaries of AE incidence in Combined Severity Grade Subsets

A brief, high-level summary of the number and percentage of participants who experienced at least 1 TEAE in the categories described below will be provided by treatment group. All deaths observed in the study will also be included in this summary.

The number and percentage of participants who experienced at least 1 TEAE will be provided and summarized by treatment group, SOC and PT, and by PT only for the following AE categories:

- TEAEs
- TEAEs (by severity)
- TEAEs with Grade 3 or higher (by severity)
- TEAEs with Grade 2 or higher
- TE treatment-related AEs
- TE treatment-related AEs with Grade 3 or higher (by severity)
- TE treatment-related AEs with Grade 2 or higher
- TE SAEs
- TE treatment-related SAEs
- TEAEs leading to premature discontinuation of study drug
- TEAEs leading to premature discontinuation of study
- TEAEs leading to death (by SOC and PT only)

Multiple events will be counted only once per participant in each summary. Adverse events will be summarized and listed first in alphabetic order of SOC, and then by PT in descending order of total frequency within each SOC. For summarizes by PT only, AEs will be summarized and listed by PT in descending order of total frequency.

In addition, data listings will be provided for the following:

- All AEs
- All SAEs
- All Deaths
- All AEs with severity of Grade 3 or higher
- All AEs leading to premature discontinuation of study drug
- All AEs leading to premature discontinuation of study

For each listing, whether the event is treatment emergent will be indicated.

## 7.1.7. Additional Analysis of Adverse Events

## 7.1.7.1. Study Drug Related Injection Site Reactions

Additional analysis of AEs will be performed for injection site reaction (ISR) related to study drug, which is defined as an AE related to study drug reported as any event within the MedDRA HLT of "Injection Site Reactions". The following summaries will be provided for each SC injection visit (eg, Day 1, Week 28) and the overall for participants in Treatment Groups 1 and 2.

- Number of participants that received SC injection(s)
- Number and percentage of participants with study drug related ISRs
- Number and percentage of participants with study drug related ISRs by grade
- Number and percentage of participants with study drug related ISRs by PT

The denominator for the percentage calculation for the by visit summary and the overall summary will be based on the total number of participants who receive at least 1 SC injection at the visit of interest and the total number of participants who receive at least 1 SC injection at any injection visit, respectively.

Duration of the ISR will also be calculated and summarized. Duration of a given ISR event is defined as the ISR stop date minus the ISR onset date plus 1 day. For ISRs with ongoing stop date, stop date will be imputed as last study date or data cut date, whichever is the earliest. Duration of ISR events in days will be summarized using descriptive statistics.

A by-participant listing for study drug-related ISRs and the corresponding duration will be provided.

#### 7.1.7.2. Study Drug Related Injection Site Induration and Nodules

Percentage of ongoing and resolved study drug related injection site induration will be summarized for each SC injection (eg, Day 15, Week 28, Week 54, etc) and the overall at both participant-level and event-level.

For the participant-level summary, if a participant had more than one injection site indurations, the participant will be counted in the "Ongoing" category unless all study drug related injection site induration events have been resolved.

For the event-level summary, duration of the resolved events will be summarized using descriptive statistics.

Study drug related injection site nodules will be summarized in the same manner as defined for study drug related injection site induration.

A by-participant listing for study drug related injection site induration and nodules and the corresponding duration will be provided.

## 7.2. Laboratory Evaluations

Laboratory data collected during the study will be analyzed and summarized using both quantitative and qualitative methods. Summaries of laboratory data will be provided for the Safety Analysis Set and will include data collected up to the last exposure date for participants who have permanently discontinued study drug, or all available data at the time of the database snapshot for participants who were ongoing at the time of an interim analysis. The analysis will be based on values reported in conventional units. When values are below the LOQ, they will be listed as such, and the closest imputed value will be used for the purpose of calculating summary statistics as specified in Section 3.7. Hemolyzed test results will not be included in the analysis, but they will be listed in by-participant laboratory listings.

#### Calcium Corrected for Albumin

Calcium corrected for albumin will be calculated and summarized for the study. The following formula will be used when both serum calcium and albumin results for a given blood drawn are available and serum albumin value is < 4.0 g/dL.

Calcium corrected for albumin (mg/dL) = serum calcium (mg/dL) +  $0.8 \times (4.0 - \text{albumin (g/dL)})$ 

Toxicity grading for calcium will be applied based on the corrected values.

#### Estimated Glomerular Filtration Rate

The following formulae will be used to calculate the estimated glomerular filtration rate using Cockcroft-Gault formula (eGFR $_{CG}$ ):

$$eGFR_{CG}$$
 (mL/min) = [(140 - age (yrs)) × weight (kg) × (0.85 if female)] / (SCr (mg/dL) × 72),

where weight is total body mass in kilograms and SCr is serum creatinine.

#### Low-Density Lipoprotein

The following formulae will be used to calculate the low-density lipoprotein (LDL) using Friedewald formula when cholesterol, high-density lipoprotein(HDL), and triglyceride for a given blood drawn are available:

LDL (mg/dL) = total cholesterol (mg/dL) – HDL (mg/dL) – triglyceride (mg/dL)/5;

The fourth generation LDL is calculated from above Friedewald formula. The third generation LDL is a direct measurement from blood drawn. Both generations of LDL will be listed in the listing. Only fourth generation LDL calculated from the Friedewald formula will be used for analysis.

A by-participant listing for laboratory test results will be provided by participant ID number and visit in chronological order for hematology, serum chemistry, and urinalysis separately. Values falling outside of the relevant reference range and/or having a severity grade of 1 or higher on the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017, will be flagged in the data listings, as appropriate.

No formal statistical testing is planned.

#### 7.2.1. Summaries of Numeric Laboratory Results

Descriptive statistics will be provided by treatment group for selected laboratory test as follows:

- Baseline values
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline laboratory value will be defined as the last measurement obtained on or prior to the date/time of first dose of study drug. Change from baseline to a postbaseline visit will be defined as the visit value minus the baseline value. The mean, median, Q1, Q3, minimum, and maximum values will be displayed to the reported number of digits; SD values will be displayed to the reported number of digits plus 1.

Median (Q1, Q3) of the change from baseline values for these selected laboratory tests will be plotted by treatment group and visit.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3.

#### 7.2.2. Graded Laboratory Values

The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 dated July 2017, will be used to assign toxicity grades (0 to 4) to laboratory results for analysis. Grade 0 includes all values that do not meet the criteria for an abnormality of at least Grade 1. For laboratory tests with criteria for both increased and decreased levels, analyses for each direction (ie, increased, decreased) will be presented separately.

For triglycerides, LDL (4th generation), and cholesterol, the toxicity grading scale is for fasting test values, so nonfasting lipid results (or lipid results without a known fasting status) will not be graded or summarized by toxicity grades.

## 7.2.2.1. Treatment-Emergent Laboratory Abnormalities

Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline visit, up to last exposure date for participants who permanently discontinued study drug, or the last available date in the database snapshot for

participants who were still on treatment at the time of an interim analysis. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment emergent.

#### 7.2.2.2. Summaries of Laboratory Abnormalities

Laboratory data that are categorical will be summarized using the number and percentage of participants in the study with the given response at baseline and each scheduled postbaseline visit.

The following summaries (number and percentage of participants) for treatment-emergent laboratory abnormalities will be provided by lab test and treatment group; participants will be categorized according to the most severe postbaseline abnormality grade for a given lab test:

- Graded laboratory abnormalities
- Grade 3 or 4 laboratory abnormalities

For all summaries of laboratory abnormalities, the denominator is the number of participants with nonmissing postbaseline values.

A by-participant listing of treatment-emergent laboratory abnormalities and treatment-emergent Grade 3 or 4 laboratory abnormalities, respectively, will be provided by participant ID number and visit in chronological order. This listing will include all test results that were collected throughout the study for the lab test of interest, with all applicable severity grades and abnormal flags displayed.

#### 7.3. Body Weight and Vital Signs

Descriptive statistics will be provided by treatment group for body weight, BMI and vital signs as follows:

- Baseline value
- Values at each postbaseline visit
- Change from baseline at each postbaseline visit

A baseline value will be defined as the last available value collected on or prior to the date/time of first dose date of study drug. Change from baseline to a postbaseline visit will be defined as the postbaseline value minus the baseline value.

In the case of multiple values in an analysis window, data will be selected for analysis as described in Section 3.8.3. No formal statistical testing is planned.
A by-participant listing of vital signs will be provided by participant ID number and visit in chronological order. Body weight, height, and BMI will be included in the vital signs listing, if space permits. If not, they will be provided separately.

#### 7.4. Prior and Concomitant Medications

Medications collected at screening and during the study will be coded using the current version of the World Health Organization (WHO) Drug dictionary. The WHO preferred name and drug code will be attached to the clinical database.

#### 7.4.1. Nonstudy Drug Antiretroviral Medications

Any nonstudy drug ARV medications are defined as any ARV medications taken prior to, during, or after the study (if collected). All nonstudy drug ARV medications will be listed. No inferential statistics will be provided.

#### 7.4.2. Concomitant Non-ARV Medications

Concomitant non-ARV medications are defined as non-ARV medications taken while a participant took study drug. Use of concomitant medications from Study Day 1 up to the last exposure date will be summarized (number and percentage of participants) by treatment group, WHO drug class and preferred name. Multiple drug use (by preferred name) will be counted only once per participant. The summary will be sorted alphabetically by drug class and then by decreasing total frequency within a class. For drugs with the same frequency, sorting will be done alphabetically.

If the start or stop date of non-ARV medications is incomplete, the month and year (or year alone, if month is not recorded) of the start or stop date will be used to determine whether the non-ARVs are concomitant or not. The medication is concomitant if the month and year of the start or stop (or year of the start or stop, if month is not recorded) of the medication does not meet either of the following criteria:

- The month and year of start of the medication is after the last exposure date
- The month and year of stop of the medication is before the first dose date of study drug

If the start and stop date of non-ARV medications are complete, the start date is not after last exposure date and the stop date is not before first dose date, or the non-ARV medications are marked as ongoing and start date is on or before last exposure date, the non-ARV medications are concomitant.

Summaries of non-ARV concomitant medications will be based on the Safety Analysis Set. No formal statistical testing is planned. A by-participant listing for all non-ARV concomitant medications will be listed and sorted by participant ID number and administration date in chronological order.

#### 7.5. Electrocardiogram Results

## 7.5.1. Investigator Electrocardiogram Assessment

The investigators' assessment of ECG results (normal; abnormal, not clinically significant; abnormal, clinically significant) are collected at screening only. A by-participant listing for ECG assessment results will be provided by participant ID number.

#### 7.6. Other Safety Measures

A data listing will be provided for participants experiencing pregnancy and participants using/misusing any substances (eg, illicit drug) during the study, respectively. Physical examination was not collected in the eCRF. Therefore, it will not be included in the analysis.

## 7.7. Participant Subgroup for Safety Endpoints

Incidence of all treatment-emergent AEs will be repeated within each subgroup defined in Section 3.4.1 using the Safety Analysis set. No formal statistical testing is planned.

#### 7.8. Changes From Protocol-Specified Safety Analysis

No change from protocol-specified safety analyses is planned.

# 8. PHARMACOKINETIC (PK) ANALYSES

#### 8.1. PK Sample Collection

Blood samples will be collected to determine PK (and metabolites, if applicable) in plasma at the following timepoints:

For Treatment Groups 1 and 2:

Plasma PK sampling will occur relative to dosing of GS-6207 at the following time points for all participants:

- Days 1, 2, and 8:
  - Predose (within 30 minutes of dosing)
  - A single timed PK sample between 1 and 6 hours postdose

- At Day 15 and at all visits with SC GS6207 injections: A single predose PK sample will be collected
- Starting at Week 4 visit, at all visits without SC GS-6207 injections: A single anytime PK sample will be collected



For Treatment Group 3:

Starting at Day 1 visit, a single anytime PK sample will be collected at all study visits.



5

For Treatment Group 4:

Starting at Day 1 visit, a single anytime PK sample will be collected at all study visits.

#### 8.2. PK Analyses Related to PK Sampling

The statistical analysis methods for the CCI

#### 8.2.1. Statistical Analysis Methods

Plasma concentration for LEN and other appropriate analytes will be listed for all participants and summarized by nominal time point for participants in the PK Analysis Set by treatment group.

Summary statistics (n, mean, 90% CI, SD, coefficient of variation [%CV], median, min, max, Q1, and Q3) will be presented for both individual participant concentration data by time point by treatment group and analyte. Moreover, the geometric mean, 95% CI, and the mean and SD of the natural log-transformed values will be presented.

The sample size for each time point will be based on the number of participants with nonmissing concentration data at that time point. The number of participants with concentration BLQ will be presented for each time point. For summary statistics, BLQ values will be treated as 0 at predose and one-half of the lower LOQ for postdose time points.

The following tables will be provided for each analyte by treatment group and visit:

Individual participant concentration data and summary statistics

The following figures may be provided for each analyte by treatment group:

- Mean (± SD) concentration data versus time (on linear and semilogarithmic scales)
- Median (Q1, Q3) concentration data versus time (on linear and semilogarithmic scales)

Individual, mean, and median postdose concentration values that are  $\leq$  LOQ will not be displayed in the figures and remaining points connected.

PK sampling details by participant, including procedures, differences in scheduled and actual draw times, and sample age will be provided in listings.

The molecular weight of TFV-DP (447.17 g/mol) and the density of 5000 million cells/mL will be used in the conversion of concentration from ng/million cells to  $\mu$ mol/L, where the value in ng/million cells \* (5000/447.17) results in the value in  $\mu$ mol/L or  $\mu$ M.

$$\frac{\textit{ng}}{\textit{million cells}} \times \frac{1 \, \textit{nmol}}{447.17 \, \textit{ng}} \times \frac{1 \, \mu \textit{mol}}{1000 \, \textit{nmol}} \times \frac{5000 \, \textit{million cells}}{1 \, \textit{mL}} \times \frac{1000 \, \textit{mL}}{\textit{L}} = \, \frac{\mu \textit{mol}}{\textit{L}} = \, \mu \textit{M}$$

### 8.2.2. Sensative Analysis

Sensitivity analysis may be conducted for the key PK analyses if the PK scientist identifies PK data as questionable or worth excluding. The sensitivity analysis will exclude specific data from analyses, if appropriate.

### 8.3. Changes From Protocol-Specified PK Analysis

No change from protocol-specified PK analyses is planned.

### 9. REFERENCES

U. S. Department of Health and Human Services, Food and Drug Administration (FDA), Center for Drug Evaluation and Research (CDER). Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment. Guidance for Industry. Silver Spring, MD. November, 2015.

## 10. SOFTWARE

SAS® Software Version 9.4. SAS Institute Inc., Cary, NC, USA.

nQuery Advisor(R) Version 7.0. Statistical Solutions, Cork, Ireland.

# 11. SAP REVISION

| Revision Date<br>(DD MMM YYYY) | Section | Summary of Revision | Reason for Revision |
|---|---|---|---|

# 12. APPENDICES

Appendix 1. Schedule of Assessments

| | Screening* | Day<br>1 <sup>b</sup> | Day 2 | CCI | Day<br>8 | Day<br>15 | Every<br>6 weeks<br>from<br>Week 4<br>to<br>Week 28<br>±2 Days | Week 38<br>±2 Days | Week 54<br>±2 Days | Week 64<br>±2 Days | Week 80<br>±2 Days | Post<br>Week 80<br>Visits <sup>e</sup><br>±6 Days | Oral<br>Bridging<br>Visits <sup>d</sup> | 30, 90,<br>180 Day<br>Follow-Up <sup>e</sup> | Early<br>Termination |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Written Informed.<br>Consent | X | | | | | | | | | | | | | | |
| Obtain demographic information | Х | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | |
| Complete Physical<br>Examination | Х | X | | | | х | X8 | | X | | х | | | | x |
| Symptom-Directed<br>Physical Examination | | | х | | Х | | Xh | X | | х | | х | х | X | |
| Vital Signs <sup>i</sup><br>(including weight) | Х | X | X | | Х | х | х | Х | Х | X | х | х | х | Х | x |
| 12-lead ECG (supine) | X | | | | | | | | | | | | | | |
| Height | X | | | | | | | | | | | | | | |
| Hematology <sup>†</sup> ,<br>Chemistry <sup>‡</sup> , Lipid<br>panel <sup>†</sup> , Urinalysis and<br>Urine Chemistry <sup>m</sup> ,<br>CD4+ Cell Count | x | x | x | | x | x | x | x | x | x | x | x | x | x | x |
| Urine Storage Sample | | X | X | | X | X | Х | X | X | X | X | X | | | х |
| Serum Pregnancy Test <sup>a</sup> | X | | | | | | | | | | | | | | X |
| Serum FSH <sup>o</sup> | X | | | | | | | | | | | | | | |
| Unine Pregnancy Test | | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| HBV, HCV Testing | X | | | | | | | | | | | | | | |
| HIV-1 Genotyping/<br>Phenotyping | X | | | | | | | | | | | | | | |
| Plasma HIV-1 RNA | X | X | X | | X | X | X | X | X | X | X | X | X | X | X |
| Plasma Storage<br>Sample | X | X | X | | X | Х | X | X | X | X | X | X | X | X | x |
| PK Plasma Collection® | | X | х | | х | X | X | X | X | X | X | X | X | | |

| | Screening* | Day<br>15 | Day<br>2 | CCI | Day<br>8 | Day<br>15 | Every<br>6 weeks<br>from<br>Week 4<br>to<br>Week 28<br>±2 Days | Week 38<br>±2 Days | Week 54<br>±2 Days | Week 64<br>±2 Days | Week 80<br>±2 Days | Post<br>Week 80<br>Visits<br>±6 Days | Oral<br>Bridging<br>Visits <sup>a</sup> | 30, 90,<br>180 Day<br>Follow-Upf | Early<br>Termination <sup>t</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CC] | | | | | | | | | | | | | | | |
| Oral GS-6207<br>Dispensation <sup>t</sup> | | X | x | | X | | х | х | X | X | х | х | х | | |
| Subcutaneous<br>GS-6207<br>Administration <sup>2</sup> | | | | | | x | х | | x | | х | x | | | |
| F/TAF Dispensation <sup>v</sup> | | X | | | | | X | X | X | X | X | X | | | |
| TAF Dispensation <sup>w</sup> | | | | | | | X | X | X | X | X | X | | | 2/1 |
| Bictegravir<br>Dispensation* | | | | | | | X | x | x | х | х | x | | | |
| B/F/TAF<br>Dispensation <sup>y</sup> | | X | | | | | X | X | x | X | | | | | |
| Study Drug<br>Accountability | | X | х | | X | X | х | x | x | х | х | X | | | |
| QoL Administration | | X | | | | X | X | | X | | X | 6<br>6 | | | |
| Injection Site Reaction<br>Assessment<br>Worksheet® | | | | | | х | х | | x | | х | | | | |
| Adverse Events/<br>Concomitant<br>Medications | х | x | x | | x | x | x | x | x | x | х | x | x | x | х |

a Screening evaluations must be completed within 30 days prior to Day 1

b Day 1 tests and procedures must be completed prior to administration of the dose of study drug. Participants must begin dosing on the same day as Day 1

c Assessments will be performed post Week 80 (Week 90, Week 106, Week 116, Week 132, Week 142) and will continue to alternate between every 10 weeks and every 16 weeks with the visit window ±6 days.

d Only applicable to participants who require oral weekly bridging if an SC injection of GS-6207 cannot be administered for any reason within the protocol visit window.

e Participants may be required to return to the clinic for a 30, 90 and 180-Day Follow-Up Visit after Early Termination visit.

f Within 72 hours of permanently discontinuing study. Counsel participant regarding the importance of continuing a complete ARV therapy in accordance to standard of care and refer participant to an appropriate HIV treatment facility.

g Complete physical exam is only required at Week 28

- h Symptom directed physical to be completed at Weeks 4, 10, 16, and 22, as necessary
- Vital signs blood pressure, pulse, respiration rate, temperature, and weight
- j Hematology: CBC with differential and platelet count
- k Chemistries: Alkaline phosphatase, AST, ALT, GGT, total bilirubin, direct and indirect bilirubin, total protein, albumin, LDH, CPK, bicarbonate, BUN, calcium, chloride, creatinine, glucose, lipase, magnesium, phosphorus, potassium, sodium, and uric acid. eGFR according to the Cockcroft-Gault formula
- 1 Fasting is not required for the lipid panel
- m Urinalysis and Urine Chemistry: including color & clarity, specific gravity, pH, glucose, ketones, bilirubin, urobilinogen, blood, nitrite, leukocyte esterase and microscopic (if microscopic elements are seen), urine protein, albumin, creatinine, phosphate, calcium, magnesium and uric acid
- n Women will have a serum test performed at Screening. Urine pregnancy test will only be done for women of childbearing potential. In Treatment Groups 1 and 2, urine pregnancy tests should be confirmed to be negative prior to subcutaneous GS-6207 administration. If any pregnancy test is positive, study drug should be immediately interrupted, and participant should come to the site for serum pregnancy test.
- o FSH test is required for women who are <54 years old and have stopped menstruating for ≥ 12 months but do not have documentation of ovarian hormonal failure.</p>
- p PK collection: For Treatment Groups 1 and 2, plasma PK sampling will occur relative to dosing of GS-6207 at Days 1, 2 and 8 predose (within 30 minutes of dosing) and a single timed PK sample between 1 and 6 hours postdose. CCI

  GS-6207, a single predose PK sample will be collected. Starting at Week 4 and at all visits without SC GS-6207, 6207 including the Oral Bridging visits, if applicable, a single anytime PK sample will be collected. PK sampling will continue at visits past Week 80.

For Treatment Groups 3 and 4 participants, starting at Day 1, a single anytime PK sample will be collected at all study visits.

- CCI
- t Treatment Group 1 and 2 oral GS-6207 lead in at Day 1, Day 2 and Day 8. Treatment Group 3 will receive oral GS-6207 lead in at Days 1 and 2 and will begin oral daily GS-6207 at Day 3.
- u Treatment Group 1 and 2 Subcutaneous administration at Day 15 and every 26 weeks
- v Treatment Group 1, 2, and 3 F/TAF once daily for 28 weeks starting at Day 1. Treatment Group 3 participants will continue F/TAF until study completion.
- w Treatment Group 1 daily oral TAF to be initiated at Week 28
- x Treatment Group 2 daily oral BIC to be initiated at Week 28
- y Treatment Group 4 daily oral B/F/TAF
- z Prior to completion of other study procedures, participants will complete HIVTSQ12, HIVDQoL, and EQ-ED-5L at Day 1 (except HIVTSQ12), Day 15 (HIVTSQ12 only), Week 4, Week 54, Week 54, Week 80. Injection Acceptability Scale and Numeric Pain Rating Scale to be completed at Day 15, Weeks 28, 54 and 80 (for Treatment Groups 1 and 2 participants only) after SC GS-6207 administration and completion of other study procedures.
- aa Provide Injection Site Reaction Assessment Worksheet and instruct the participants to measure and report injection site reactions following the administration of the subcutaneous injections (for Treatment Group 1 and 2 participants only)

### Appendix 2. Programming Specification

1) If the age from the Day 1 eCRF is not available, age will be calculated as follows:

Only year is provided for the date of birth (DOB). Use July 1 for the month and day.

- a) AGE (years) is calculated from the number of days between the DOB and Study Day 1,
- Use the SAS INTCK function to determine the number of "1st-of-month days" (eg, January 1st, February 1st, March 1st) between DOB and Day 1 (inclusive),
- c) Divide the result in (b) by 12,

AGE = the integer of the result in (c),

Age for laboratory test reference range will be based on the age at the sample collection date.

- 2) All screened participants refer to all participants who are screened (ie, with non-missing screening date) and have a screening number. For summaries the same participant is counted only once.
- Screen failure participants are the participants who were screened and answered "No" for any inclusion criteria or "Yes" for any exclusion criteria regardless of which version of protocol the participant was consent to.
- 4) Participants in the randomized analysis set are defined as participants randomized into the study. IXRSRAND is the source to determine whether the participant is randomized (ie, participant with non-missing RGMNDTN in the IXRSRAND dataset), and confirmed by the eCRF ENROLL dataset (ie, ENROLLYN = "Yes" in ENROLL dataset).
- 5) Randomized treatment (ie, TRT01P in ADSL) is derived from IXRSRAND, while actual treatment received (ie, TRT01A in ADSL) is assigned as the randomized treatment if participant took at least 1 dose of study drug and assigned as blank if the participant was never dosed.
- 6) In the disposition table, the reasons for premature discontinuation are displayed in the order as they appear on the eCRF.
- 7) Body mass index (BMI)

BMI will be calculated only at baseline as follows:

— BMI = (weight [kg]) / (height [meters]<sup>2</sup>)

Baseline height and weight will be used for this calculation if available.

SAS codes for the treatment comparison for demographics and baseline characteristics tables.

CMH test for nominal variable (Y), the p-value from the general association test should be used for nominal variables:

```
proc freq;
tables trt * Y /cmh; /*general association test*/
run:
```

CMH test for ordinal variable (Y), the p-value from the row mean score test should be used for ordinal variables:

```
proc freq;
tables trt * Y / cmh2 ; /*row mean score test*/
run;
```

Kruskal-Wallis test for continuous variable (Y):

```
proc nparlway wilcoxon;
class trt;
var Y;
run;
```

- For race and ethnicity, "Not Permitted", "Missing", or "Other" will be excluded from percentage calculation and also excluded for p-value generation for categorical data analysis (eg, CMH test or Kruskal-Wallis test).
- Study Day 1, Last Dose Date and Last Exposure Date
  - a) All the key dates were defined in Section 3.8.1.
- 11) Study Day 1 and Last Dose Date
  - a) All the key dates were defined in Section 3.8.1.
  - Study Day 1 is defined as the earliest of the dose start dates from any Study Drug Administration eCRF (ie, EX, EX\_ARV or EX\_IV).
  - c) Last Dose Date is defined for participants who prematurely discontinued study drug in Treatment Groups 1 to 3, or completed study drug at main phase in Treatment Group 4 according to Study Drug Completion eCRF(ie, SDRGCOMP).
    - i) For participants who receive SC injection(ie, A participant has data in EX\_IV.) and took any oral bridging LEN(ie, A participant has data in EX.EXTRT="Oral GS-6207" and EX. EXDOSFRQ\_STD="1TIMEPERWEEK"), the last dose date is defined as earliest of the last dose date of oral bridging LEN(ie, the last dose date of EX.EXTRT="Oral GS-6207" and EX. EXDOSFRQ\_STD="1TIMEPERWEEK") or oral QD drug(ie, the last dose date in EX\_ARV),

- ii) For participants who receive SC injection(ie, A participant has data in EX\_IV.) and did not take any oral bridging LEN, the last dose date is defined as the latest nonmissing end date of the study drug used with LEN (ie, the last dose date in EX\_ARV).
- iii) For participants who do not receive SC injection(ie, A participant has no data in EX\_IV.), the last dose date is defined as the earliest of the last dose date of any study drug (ie, the earliest of last dose date in EX or EX\_ARV).
- d) Study drug administration: Oral reload will be recorded as an "Unscheduled" visit in the Study Drug Administration eCRF. Participants with oral reload prior to the 1st dose of SC have "Unscheduled" dosing visits occurred prior to Day 15 visit. Participants who received a total of 5 tablets of LEN (300 mg) (ie, 2 x 300 mg LEN tablets each for the first 2 days and 1 x 300 mg LEN tablet on the 8th day) prior to "Unscheduled" dosing visits followed by Day 15 visit will be classified as oral reload due to missing scheduled SC dosing. Otherwise, participants will be classified as oral reload due to missing scheduled oral dosing visit.
- 12) Adherence to QD Study Drug(s): (excluding oral lead-in LEN and oral bridging LEN)
- a) Adherence based on 1 study drug(Treatment Groups 1, 2, and 4):

Adherence (%) = 
$$100 \times \frac{Total \text{ No. of pills taken}}{Total \text{ No. of pills prescribed}}$$
  
 $\Sigma \text{ No. of pills taken at each dispensing period for each study drug}$ 

 $= 100 \times \frac{\sum \text{No. of pills taken at each dispensing period for each study } \text{drug}^{[1]}}{\sum \text{No. of pills prescribed at each dispensing period for each study } \text{drug}^{[2]}}$ 

b) Adherence based on 2 study drugs(Treatment Group 3):

$$Adherence(\%) = 100 \times \frac{Total \, No. of \, pills \, taken}{Total \, No. of \, pills \, prescribed}$$

$$= 100 \times \frac{\sum \sum No. of \, pills \, taken \, at \, each \, dispensing period \, for \, each \, drug^{[1]}}{\sum \sum No. of \, pills \, prescribed at \, each \, dispensing period \, for \, each \, drug^{[2]}}$$

#### 13) Efficacy Analysis

a) For categorical efficacy response (eg, Participants with HIV-1 RNA < 50 copies/mL as determined by US FDA-defined snapshot algorithm, M=F, or M=E Analyses): the proportion difference between LEN-containing regimen groups (Treatment Groups 1 to 3) and the B/F/TAF group (Treatment Group 4) and its 95% CIs are calculated based on the MH proportion adjusted by baseline HIV-1 RNA stratum (≤ 100,000 vs. > 100,000 copies/mL) (see SAP Section 6.2 and Section 6.3 for details). The following SAS code will be used to compute p-value, where brnac is the baseline HIV-1 RNA stratum, trtgrp is the treatment, and response is the categorical efficacy response.

```
proc freq data=adeff;
   tables brnac*trtgrp*response/cmh; /*p value from general
   association*/
run;
```

b) All the ANOVA model for continuous efficacy variable (eg, CD4+): The differences in changes from baseline in log<sub>10</sub> HIV-1 RNA and CD4+ cell count between treatment groups and the associated 95% CI will be constructed using an ANOVA, including baseline HIV-1 RNA stratum brnac, region stratum region, and treatment trtgrp as fixed effects in the model.

```
proc glm data=adeff;
   class brnac region trtgrp;
   model CD4=brnac region trtgrp;
   lsmeans trtgrp /alpha=0.05 cl pdiff;
run;
```

# GS-US-200-4334-Final-SAP-v1.0

# **ELECTRONIC SIGNATURES**

| Signed by | Meaning of Signature | Server Date<br>(dd-MMM-<br>yyyy hh:mm:ss) |
|---|---|---|
| PPD | Biostatistics eSigned | 18-Jan-2024<br>04:31:32 |
| PPD | Clinical Pharmacology<br>eSigned | 18-Jan-2024<br>22:50:23 |
| PPD | Clinical Development eSigned | 18-Jan-2024<br>23:08:08 |